CLINICAL TRIAL: NCT06681116
Title: Use of Nanotechnology Structured Water for the Prevention of Recurrent Stone Formation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ALI KAMAL M. SAMI (Other)
Responsible Party: Sponsor-Investigator, ALI KAMAL M. SAMI, Lecturer, College of Medicine,, University of Sulaimani
Organization: University of Sulaimani (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 173
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Renal Stones; Idiopathic Hypercalciuria
Keywords: recurrent renal stones; idiopathic hypercalciuria; nano-water; hydrochlorthiazide
MeSH Terms: conditions — Nephrolithiasis | interventions — Hydrochlorothiazide

STUDY DESIGN:
Intervention Model Description: Three groups that run parallel and receive the different allocated modalities and are followed up for three consecutive years
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: neither the participants nor the investigators or the care givers and the outcome assessors knew the group of patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with idiopathic hypercalciuria Group A (Experimental): Patients receiving nano-water in a daily dose of 20 mL/Kg
  Interventions: Dietary Supplement: structured nano-water
- Patients with idiopathic hypercalciuria Group B (Active Comparator): Patients receiving Hydrochlorothiazide in a daily dose of 50 mg.
  Interventions: Drug: Hydrochlorothiazide (HCTZ)
- Patients with idiopathic hypercalciuria Group C (Placebo Comparator): Patients receiving ordinary bottled drinking water in a daily dose of 20 mL/Kg
  Interventions: Other: ordinary bottled drinking water

INTERVENTIONS:
Dietary Supplement: structured nano-water — Hydrochlorothiazide is a drug used to prevent recurrent renal stone formation in patients with idiopathic hypercalciuria
  Arms: Patients with idiopathic hypercalciuria Group A
Drug: Hydrochlorothiazide (HCTZ) — hydrochlorothiazide is a drug used to prevent recurrent stone formation i patients with idiopathic hypercalciuria
  Arms: Patients with idiopathic hypercalciuria Group B
Other: ordinary bottled drinking water — Patients with idiopathic hypercalciuria receiving regular bottled drinking water as a placebo to see its effect.
  Arms: Patients with idiopathic hypercalciuria Group C

SUMMARY:
We assessed the effect of structured nano-water in the prevention of recurrent stone formation in patients with recurrent calcium oxalate stones and hypercalciuria.

DETAILED DESCRIPTION:
The majority of stones (85%) contain primarily calcium oxalate. Most renal stones are idiopathic calcium stones, and the most common predisposing factor in these patients is hypercalciuria. Structured nano-water is a new type of water that has been prepared using different types of energy fields electromagnetic fields to produce this structured nano- water that has new and different characteristics from the ordinary water.

In this study, we compared the efficacy of the nano- water with hydrochlorothiazide and with ordinary bottled drinking water in the prevention of recurrent renal stones in patients with idiopathic hypercalciuria.

We conducted a three-year randomized trial comparing the effect of structured water with the effect of hydrochlorothiazide and ordinary bottled water in 325 patients with recurrent calcium oxalate stones and hypercalciuria.

The patients were randomly divided into three groups. Group A included 108 patients who used structured nano-water in a dose of 20 mL/kg as a daily dose.

Group B of 107 patients used 50 mg hydrochlorothiazide tablets as a daily dose, and group C consisted of another 110 patients used ordinary drinking bottled water in a daily dose of 20 mL/kg .

The assessments were done by urine analysis with renal ultrasonography and radiology ( Kidney Ureter Bladder KUB X-rays) were done at baseline, at yearly intervals, also at any time of recurrence, and at the end of the 3 years (36th month).

The patients, care providers, and the investigators were blinded about the type of water used since the water bottles were unlabeled when given to the patients.

All patients were informed and signed a written informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic hypercalciuria
* history of previous renal stones

Exclusion Criteria:

* already present renal stones
* previous surgery of the kidneys
* Congenital anomalies of the urinary system
* Renal failure
* Allergy to hydrochlorothiazide

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2015-02-16 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
Recurrent renal stones | From enrollment to the end of treatment at 36 months
  recurrent renal stone were diagnosed by ultrasound and X-ray ( kidney ureter Bladder X-ray)

CONTACTS AND LOCATIONS:
Overall Officials: Ali K M. Sami, MBChB FIBMS, Principal Investigator — College of Medicine, University of Sulaimani
Locations (1):
- College of Medicine, University of Suliamani, Sulaymaniyah, Kurdistan Region, Iraq

IPD SHARING:
Plan to Share IPD: No
Patients agreed to participate in this clinical trial based on keeping confidentiality about their personal informations